CLINICAL TRIAL: NCT01485094
Title: Evaluation of the Efficacy, Tolerability, and Safety of 7 Days of Treatment With GRT6010 or Pregabalin in Comparison to Placebo in Subjects With Peripheral Neuropathic Pain.
Brief Title: A Study to Assess the Safety and Efficacy of 7 Days Treatment With a Novel Analgesic in Subjects With Peripheral Neuropathic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was early terminated after it was concluded that there was no added benefit from exposing further participants after an unblinded interim analysis.
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 967165; 2011-002092-42 (EudraCT Number)
Record Dates: First submitted 2011-10-05; First posted 2011-12-05 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Neuralgia
Keywords: neuralgia; postherpetic
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Matching placebo (Placebo Comparator): Oral administration. Pain not sufficiently controlled may be treated with acetaminophen.
  Interventions: Drug: Matching Placebo
- GRT6010 (Experimental): Oral administration. Pain not sufficiently controlled may be treated with acetaminophen.
  Interventions: Drug: GRT6010
- Pregabalin (Active Comparator): Oral administration. Pain not sufficiently controlled may be treated with acetaminophen.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: GRT6010 — Oral solution given once daily.
  Arms: GRT6010
Drug: Pregabalin — Over-encapsulated pregabalin capsules 75mg twice daily on Days 1 to 3, and 150mg twice daily on Days 4 to 7.
  Other Names: Lyrica®
  Arms: Pregabalin
Drug: Matching Placebo — Matching Placebo capsules to the over-encapsulated Pregabalin capsules and Matching Placebo oral solution to the GRT6010 solution.
  Capsules twice daily on Days 1 to 7. Solution once daily.
  Arms: Matching placebo

SUMMARY:
The purpose of this trial is to determine whether a novel analgesic is effective in treating of neuropathic pain caused by herpetic infection, surgery, or trauma.

DETAILED DESCRIPTION:
This trial evaluates the effectiveness of a novel analgesic in peripheral neuropathic pain in a mixed patient population. Participants were treated for one week and randomly assigned to the novel analgesic, pregabalin, or placebo. Pain will be characterized before and at the end of this period. This trial required the participants to stay at the investigational site for 14 consecutive days.

The enrollment visit took place Day -28 to Day -16. Participants tapered down their existing medication from Visit 2 (Day -17 to Day -5) to Visit 3 and were given rescue medication (paracetamol/acetaminophen). At Visit 3 participants were hospitalized (Day -4). The baseline evaluation period took place from Day -3 to Day -1. Randomization to one of the three treatment arms was possible after the last assessment on Day - 1 alternatively randomization took place on Day 1. This was followed by the double-blind treatment period (Day 1 to Day 7). The participants were follow-up thereafter up to day 36 (Day 34 to 38). Participants were permitted to resume their previous medication.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to 75 years
* Presence of persistent neuropathic pain for at least 6 months at the time of the Enrollment Visit. Allowed reasons for neuropathic pain are: modified radical mastectomy, breast conserving surgery, or cosmetic breast surgery. [Germany: subjects after cosmetic breast surgery may not be enrolled.]
* Presence of "probable" or "definite" neuropathic pain.
* Presence of dynamic mechanical allodynia on the affected side, or alternatively, the mechanical pain sensitivity for any of the pinprick stimuli is higher on the affected compared to the contralateral side.
* At either Visit 5 or Visit 6: Presence of an average evoked pain intensity score of >20 on the 0 100 point numeric rating scale (NRS) for at least 1 of the 3 clinical sub-tests for dynamic mechanical allodynia (i.e., standardized brush, cotton wool tip or cotton wisp). The average will be calculated as the arithmetic mean of all measurements per sub test. Alternatively, the arithmetic mean of the 5 test replicates for any of the pinprick stimuli for mechanical pain sensitivity is at least 3 times higher for the affected side compared to the contralateral side.
* Presence of an average ongoing pain intensity score of >4 to <9 on the 0-10 point numerical rating scale (NRS) without the use of rescue medication within the 3 day Baseline pain intensity evaluation Period with at least 7 of 9 assessments being present.
* Dissatisfaction with the current treatment (i.e., lack of efficacy or intolerable side effects) if taking an opioid or non opioid analgesic medication for the painful neuropathy before enrollment.

Exclusion Criteria:

* Any kind of hepatic impairment at Visit 1 or at Visit 3.
* Either active hepatitis within the past 3 months or presence of chronic hepatitis irrespective of its activity status.
* Estimated creatinine clearance of less than 60 mL/minute x 1.73 m2 at either Visit 1 or at Visit 3.
* Clinically relevant cardiac disease (e.g., unstable angina pectoris, angina pectoris Canadian Cardiovascular Society [CCS] Grade III to IV, acute myocardial infarction within the last 3 months, cardiac insufficiency New York Heart Association [NYHA] Class III to IV).
* Electrocardiogram (ECG) with clinically relevant findings at either Visit 1 or at Visit 3, including but not limited to repeated prolongation of QTc > 450 ms (Fridericia correction), or a history of additional risk factors for torsade de pointes (e.g., family history of Long QT Syndrome).
* Clinically relevant pulmonary disease (e.g., Medical Research Council breathlessness scale of 2 or above).
* Specific antitumor therapy within the last 6 months, e.g., adjuvant radiotherapy or chemotherapy, biologics, or angiogenesis inhibitors.
* CYP2D6 poor metabolizer phenotype as predicted by CYP2D6 genotyping.
* Presence of confounding pain conditions (e.g., ulnar nerve entrapment, radial nerve injury associated with major soft-tissue or bone damage, cervico-thoracic radiculopathy, carpal tunnel syndrome, chemotherapy-induced peripheral neuropathy, or complex regional pain syndrome type I or type II).
* Phantom breast or phantom limb pain.
* Presence of exclusively negative symptoms of neuropathic pain (e.g., hypoesthesia or total anesthesia) in the affected area.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Trials, Study Director — Grünenthal GmbH
Locations (12):
- Germany (2):
  - DEU001, Mainz
  - DEU002, Regensburg
- Hungary (4):
  - HUN004, Esztergom
  - HUN003, Győr
  - HUN001, Miskolc
  - HUN008, Szikszó
- Poland (3):
  - POL002, Gdansk
  - POL004, Lublin
  - POL005, Warsaw
- United Kingdom (3):
  - GBR003, Belfast
  - GBR001, Glasgow
  - GBR002, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on the 23 Feb 2012 and the last participant completed the trial on the 18 Jan 2013. A decision to terminate the trial was taken on 18 Dec 2012 after the results of an interim analysis.
Pre-assignment Details: 114 participants signed informed consent to participate in the trial. 59 participants of the planned 90 were randomized and 57 received study drug (investigational medicinal product).
Groups:
- Matching Placebo: Oral administration. Pain not sufficiently controlled may be treated with acetaminophen.
  Matching Placebo: Matching Placebo capsules to the over-encapsulated pregabalin tablets and Matching Placebo oral solution to the GRT6010 solution.
  Capsules twice daily on Days 1 to 7. Solution once daily.
- Pregabalin: Oral administration. Pain not sufficiently controlled may be treated with acetaminophen.
  Pregabalin: Over-encapsulated Pregabalin tablets 75mg twice daily on Days 1 to 3, and 150mg twice daily on Days 4 to 7.
Period: Overall Study
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Started | 20 | 20 | 19
Completed | 17 | 18 | 18
Not Completed | 3 | 2 | 1
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat
Groups:
- Matching Placebo: Oral administration. Pain not sufficiently controlled may be treated with acetaminophen.
  Matching Placebo to the over-encapsulated pregabalin tablets and Matching Placebo oral solution to the GRT6010 solution.
  Capsules twice daily on Days 1 to 7. Solution once daily.
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | GRT6010 | Pregabalin | Total
Number analyzed (Participants) | 19 | 19 | 19 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 16 | 15 | 49
  >=65 years | 1 | 3 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.53 (14.83) | 54.00 (9.93) | 50.53 (14.55) | 50.35 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 12 | 35
  Male | 7 | 8 | 7 | 22
Region of Enrollment [Number; unit: participants]
  Hungary | 3 | 2 | 2 | 7
  Poland | 0 | 1 | 0 | 1
  Germany | 1 | 1 | 1 | 3
  United Kingdom | 15 | 15 | 16 | 46
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 27.56 (3.80) | 27.37 (3.03) | 27.27 (3.32) | 27.40 (3.34)
Time since diagnosis of neuropathic pain [Mean (Standard Deviation); unit: months] | 32.95 (27.84) | 83.26 (49.86) | 63.32 (54.79) | 59.84 (49.49)

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Baseline and End-of-double-blind Treatment Ongoing Pain Intensity Scores
Description: The baseline pain intensity score was calculated as a mean of pain intensity scores during the Baseline Period (from Day -3 to Day -1). The ongoing pain intensity data from Day-3 to Day 7 was used. For the analysis, only pain scores on days where participants received study drug were considered. The primary efficacy analysis of the ongoing pain intensity score were analyzed in a Bayesian framework, via a mono exponential decay model, with the baseline Numeric Rating Score (NRS) as intercept. Considering the inclusion criteria of baseline pain intensity being in the range from 4 to 9, the range in ongoing pain intensity difference between baseline and end-of-double-blind treatment can be from 6 (worst possible value) to -9 (best possible value). A negative value indicates improvement whilst on the treatment.
Time Frame: Baseline; Day 7 (end of double blind treatment)
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- GRT6010: Oral administration. Pain not sufficiently controlled may be dosed with acetaminophen.
  GRT6010: Oral solution given once daily.
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 19 | 19 | 19
units on a scale | -2.55 (2.15) | -2.30 (1.73) | -2.33 (1.58)

2. Primary Outcome: The Difference Between Baseline and End-of-double-blind Treatment Brush-evoked Pain Intensity Scores
Description: The difference between baseline and end-of-double-blind treatment brush-evoked pain intensity scores compared to placebo on a 0-100 point NRS (measured as part of the dynamic mechanical allodynia assessments).
  Each participant rated each brush-evoked pain intensity on a 0 to 100 point Numerical Pain Rating Scale, with 0 indicating 'No Pain' and 100 indicating 'most intense pain imaginable'. Lower values compared to an individual subject's baseline are an improvement in symptoms.
  The baseline brush-evoked pain intensity score was defined as the average of the geometric mean of all of the values obtained on Day -2 and Day -1, and compared with the scores obtained on day 6 and 7.
  For the analysis, only pain scores on days where participants received study drug were considered.
  A negative change indicates a decrease in brush-evoked pain intensity from baseline.
Time Frame: Baseline and day 7 (end of double blind treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 19 | 19 | 19
units on a scale | -11.17 (15.88) | -14.31 (20.90) | -9.79 (13.69)

3. Secondary Outcome: Assessment of Responder Rates
Description: The assessment was performed on Day 7.
  The percentage of change from baseline (Day -3 to Day -1, i.e. the 3 days in the days prior to first dose) in the daily ongoing pain intensity was calculated at Day 7.
  The percentage of change from baseline in the daily ongoing pain intensity was calculated at Day 7 as follows:
  % change = (Baseline Pain Intensity - Daily pain intensity at treatment visit) / Baseline Pain Intensity × 100
  The threshold values represent an improvement in ongoing pain intensity greater than 20, 30, 40, 50, 60, 70, 80 or 90% as per calculation.
  Participants who showed a worsening in their daily pain intensity or who prematurely discontinued the trial were regarded as non-responders in terms of the respective treatment.
Time Frame: Day 7 (end of double blind treatment)
Measure: Number; unit: participants
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 19 | 19 | 19
participants
  20% Threshold | 12 | 14 | 13
  30% Threshold | 11 | 10 | 8
  40% Threshold | 8 | 9 | 6
  50% Threshold | 5 | 7 | 4
  60% Threshold | 4 | 4 | 4
  70% Threshold | 4 | 1 | 2
  80% Threshold | 3 | 0 | 2
  90% Threshold | 1 | 0 | 2

4. Secondary Outcome: Onset of Current Pain Relief
Description: Onset of current pain relief defined as the first time-point at which the participant reports a decrease of a 1-point reduction in current pain relative to baseline (day -3 to day -1), after start of treatment with study drug on Day 1.
  Due to the early termination of the trial this analysis was not performed.
Time Frame: Day 1 to Day 7 (end of double blind treatment)
Population: Due to the early termination of the trial this analysis was not performed.
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Onset of Ongoing Pain Relief
Description: Onset of ongoing pain relief defined as the first time-point at which the participant reports a decrease of more than 1-point reduction in ongoing pain relative to baseline (day -3 to day -1), after start of treatment with study drug on Day 1. Study drug intake started on Day 1.
  Due to the early termination of the trial this analysis was not performed.
Time Frame: Day 1 to Day 7 (end of double blind treatment)
Population: Due to the early termination of the trial this analysis was not performed.
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in Neuropathic Pain Symptom Inventory Scores on Day 7 From Baseline (Day -1)
Description: The Neuropathic Pain Symptom Inventory (NPSI) Score is an assessment of neuropathic pain symptoms.
  A participant answered 10 questions on an 11-point scale 0 (no pain) to 10 (most intense pain imaginable).
  The total NPSI score is the sum of all ten responses and ranges between 0 and 100.
  The baseline score and the mean NPSI change is reported over the double-blind treatment period. A negative mean change in score on Day 7 indicates an improvement on this 0 to 100 point scale from baseline for the total score.
  For pain descriptions burning, pressing, paroxysmal (pain like electric shocks or stabbing), evoked (due to touch) and paresthesia (sensation that is not unpleasant) or dysesthesia (unpleasant) subscores a negative mean change indicate an improvement on the 11 point scale. A participant will score 10 to indicates the worst imaginable symptom, e.g. worst burning imaginable. A participant will score 0 if there is no burning, i.e. the symptom is absent.
Time Frame: Day -1; Day 7 (end of double blind treatment)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 19 | 19 | 19
units on a scale
  Day -1 Baseline NPSI total score | 59.11 (16.47) | 58.05 (16.75) | 55.84 (22.97)
  Day 7 Change in NPSI total score | -23.89 (18.81) | -18.95 (19.56) | -16.79 (25.31)
  Day -1 Baseline Burning spontaneous pain | 5.79 (1.87) | 5.68 (2.36) | 5.63 (3.06)
  Day 7 Change in burning spontaneous pain | -2.53 (2.34) | -1.58 (2.32) | -2.0 (2.03)
  Day -1 Baseline pressing spontaneous pain | 4.47 (2.54) | 4.97 (3.07) | 4.45 (2.91)
  Day 7 Change in pressing spontaneous pain | -1.74 (2.31) | -1.68 (1.88) | -0.58 (2.58)
  Day -1 Baseline paroxysmal pain | 6.39 (2.07) | 6.03 (2.2) | 6.76 (2.39)
  Day 7 Change in paroxysmal pain | -2.92 (2.21) | -1.82 (2.7) | -2.26 (2.84)
  Day -1 Baseline evoked pain | 6.02 (2.06) | 5.83 (1.94) | 5.67 (2.31)
  Day 7 Change in evoked pain | -2.16 (2.30) | -2.03 (2.22) | -2.05 (2.89)
  Day -1 Baseline paresthesia or dysesthesia | 6.76 (2.12) | 6.45 (1.79) | 5.39 (3.18)
  Day 7 Change in paresthesia or dysesthesia | -2.79 (2.28) | -2.13 (1.94) | -1.47 (3.25)

7. Secondary Outcome: Difference in Patient's Global Impression of Change
Description: In the Patient Global Impression of Change (PGIC) the participant indicates the perceived change over the 7 day treatment period. The participant is requested to choose one of seven categories. Scores range from very much improved to very much worse.
Time Frame: Day 7 (end of double blind treatment)
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 19 | 19 | 19
participants
  Very much improved | 5 | 2 | 5
  Much improved | 4 | 6 | 4
  Minimally improved | 5 | 8 | 8
  No change | 5 | 2 | 1
  Minimally worse | 0 | 1 | 0
  Much worse | 0 | 0 | 1
  Very much worse | 0 | 0 | 0

8. Secondary Outcome: The Difference Between Baseline and End-of-double-blind Treatment Scores for Dynamic Mechanical Allodynia and Mechanical Pain Sensitivity Compared to Placebo
Description: Allodynia is pain due to a stimulus that does not normally provoke pain. Dynamic mechanical allodynia was assessed using a set of 3 light tactile stimulators as moving innocuous stimuli.
  Each participant gave numerical pain ratings for each of 15 stimuli at the affected side.
  Mechanical pain sensitivity was assessed using a set of 7 weighted pinprick stimuli to obtain the stimulus-response function for pinprick-evoked pain.
  The participant gave a numerical pain ratings for each of 35 pinprick stimuli at the affected site.
  Dynamic mechanical allodynia and mechanical pain sensitivity was calculated as the geometric mean of all numerical ratings. The values obtained on Day -2 and -1 were taken as the baseline and values on Day 6 and 7 were taken as the end of treatment. A negative change indicates an improvement on the 0 (no pain) to 100 point scale, where 100 indicates the worst imaginable pain.
Time Frame: Day 7 (end of double blind treatment)
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 19 | 19 | 19
units on a scale
  Mechanical pain sensitivity (Affected side) | -12.26 (23.28) | -14.60 (17.79) | -13.86 (15.32)
  Dynamic mechanical allodynia (Affected side) | -11.12 (17.49) | -13.81 (19.81) | -9.63 (13.00)

9. Secondary Outcome: Change in Area of Static Allodynia and Dynamic Allodynia From Baseline
Description: Allodynia is pain due to a stimulus that does not normally provoke pain. To measure the areas of dynamic and static allodynia, a point lying in the center of the area of maximum pain was marked at baseline (Day -2 and -1). From the baseline point, 8 radii were drawn.
  The area of dynamic allodynia was determined by gently stroking the skin with a standardized brush along the lines. The participant was asked to report when the sensation became unpleasant.
  The area of static allodynia was determined by a 128 mN (millinewton) pinprick stimulus along the lines of the 8 radii while asking the subject to report when the sensation became unpleasant.
  The area was calculated from the summing of the 8 triangles that are generated from the points along each of the 8 radii at which unpleasantness was reported. The larger the area in square centimeters the more allodynia. A reduction in the area of allodynia indicates improvement.
Time Frame: Baseline; Day 7 (end of double blind treatment)
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 19 | 19 | 19
square centimeters
  Dynamic allodynia area at baseline | 154.79 (190.33) | 152.11 (178.43) | 98.4 (99.20)
  Change in area of dynamic allodynia | 11.36 (153.96) | -73.98 (149.54) | -32.78 (75.96)
  Static allodynia area at baseline | 352.97 (443.83) | 286.21 (264.05) | 244.75 (250.03)
  Change in area of static allodynia | -58.01 (415.29) | -137.47 (234.46) | -95.16 (108.04)

10. Secondary Outcome: Difference in Leeds Sleep Evaluation Questionnaire After 7 Days of Treatment
Description: On the last day of the double-blind treatment period sleep was evaluated using the Leeds sleep evaluation questionnaire. This questionnaire has 10 self-rating 100 mm line analogue questions concerning sleep and early morning behavior. The higher the score, i.e. the closer the value is to 100 the worse the rating by the participant.
  The 10 responses are grouped into 4 subscores:
  * The ease of getting to sleep.
  * The perceived quality of sleep.
  * The ease of awakening from sleep.
  * The integrity of behavior following wakefulness.
Time Frame: Day 7
Population: Intention-to-treat. No responses were obtained from 2 participants, one in the placebo and one in the pregabalin treatment arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 19 | 19 | 19
units on a scale
  Day 7 ease of getting to sleep | 36.37 (14.77) | 41.25 (14.77) | 32.57 (22.81)
  Day 7 perceived quality of sleep | 42.69 (19.73) | 42.33 (23.01) | 37.06 (24.86)
  Day 7 ease of awakening from sleep | 44.94 (21.04) | 48.29 (17.51) | 46.56 (21.29)
  Day 7 integrity of behavior following wakefulness | 46.91 (22.55) | 44.88 (23.97) | 44.35 (17.35)

11. Secondary Outcome: Change in painDETECT Grading From Baseline (Day -1) to End of Double-blind Treatment (Day 7)
Description: The painDETECT questionnaire was used to determine the possibility of the presence of a neuropathic pain component. It is a participant completed questionnaire. A total score is calculated between 0 and 38 for each participant. Participants with a score between 0 and 12 are graded as "negative" and having "no neuropathic pain component". Scores between 19 and 38 result in a "positive" grading, in other words having "presence of neuropathic component". Values from 13 to 18 result in participants being graded as having an "unclear" neuropathic component to their pain. The painDETECT questionnaire was first administered on Day-1 (baseline). The data reported is for before treatment start (Day -1) and the change from baseline on Day 7 (end of the double-blind period).
Time Frame: Day 7 (end of double blind treatment)
Population: Intent-to-treat. 5 participants did not complete the painDETECT questionnaire on Day 7. Two participants in both the placebo and pregabalin treatment arm and 1 in the GRT6010 treatment arm.
Measure: Number; unit: participants
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 19 | 19 | 19
participants
  Day -1 no neuropathic pain component | 0 | 0 | 0
  Day 7 no neuropathic pain component | 1 | 2 | 2
  Day -1 Unclear neuropathic component | 2 | 1 | 5
  Day 7 Unclear neuropathic component | 4 | 4 | 3
  Day -1 Presence of neuropathic component | 17 | 18 | 14
  Day 7 Presence of neuropathic component | 12 | 12 | 12

12. Secondary Outcome: Daily Current Pain Intensity
Description: Participants recorded their current pain intensity score 3 times a day, using a 0 -10 (11 point) Numeric Rating Scale where a rating of 0 corresponded to "No Pain" and a rating of 10 to "Pain as bad as you can imagine".
  The daily current pain intensity reported was derived as the mean of the 3 current pain intensity assessments taken on the day from all participants in the treatment group.
  The lower the value on the 11 point scale the less pain was reported on a treatment.
Time Frame: Baseline; Day 10
Population: Intent-to-Treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Number analyzed (Participants) | 19 | 19 | 19
units on a scale
  Baseline | 6.32 (1.72) | 6.52 (0.98) | 6.13 (1.49)
  Day 1 | 4.82 (2.17) | 5.74 (1.47) | 5.37 (1.86)
  Day 2 | 4.49 (2.34) | 5.19 (2.02) | 4.58 (1.97)
  Day 3 | 4.46 (2.19) | 4.68 (1.77) | 4.61 (1.93)
  Day 4 | 4.09 (2.50) | 4.75 (1.92) | 4.47 (1.93)
  Day 5 | 3.82 (2.36) | 4.61 (2.04) | 3.95 (1.78)
  Day 6 | 4.13 (2.43) | 4.16 (1.81) | 4.08 (1.85)
  Day 7 | 3.64 (2.41) | 3.84 (1.82) | 3.63 (2.06)
  Day 8 | 3.68 (2.09) | 3.76 (1.81) | 3.85 (2.14)
  Day 9 | 4.21 (2.30) | 4.28 (1.88) | 4.05 (2.32)
  Day 10 | 4.06 (2.35) | 4.35 (1.88) | 4.15 (2.47)

ADVERSE EVENTS:
Groups:
- Matching Placebo: Oral administration. Pain not sufficiently controlled may be dosed with acetaminophen.
  Matching Placebo: Matching Placebo capsules to the Pregabalin capsules and Matching Placebo oral solution to the GRT6010 solution.
  Capsules twice daily on Days 1 to 7. Solution once daily.
- Pregabalin: Oral administration. Pain not sufficiently controlled may be dosed with acetaminophen.
  Pregabalin: Pregabalin capsules 75mg twice daily on Days 1 to 3, and 150mg twice daily on Days 4 to 7.
Arm/Group | Matching Placebo | GRT6010 | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 16/19 | 16/19 | 17/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo (N=19) | GRT6010 (N=19) | Pregabalin (N=19)
Headache (Nervous system disorders) | 8 | 4 | 9
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 4
Fatigue (General disorders) | 5 | 3 | 3
Dizziness (Nervous system disorders) | 7 | 3 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Hot flush (Vascular disorders) | 0 | 2 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Local reaction (General disorders) | 0 | 1 | 0
Puncture site reaction (General disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Balance disorder (Nervous system disorders) | 1 | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Somnolence (Nervous system disorders) | 3 | 0 | 3
Tremor (Nervous system disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Catheter site pain (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1
Feeling drunk (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Infected naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Depersonalisation (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Sleep talking (Psychiatric disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Mole excision (Surgical and medical procedures) | 1 | 0 | 0
Infusion Site Pain (General disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Joint publications are only possible if both parties agree. All editorial decisions will be jointly taken by the sponsor and the international coordinating investigator. The sponsor reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.